CLINICAL TRIAL: NCT02142218
Title: Expanded Access Program With Nivolumab for Subjects With Histologically Confirmed Stage III (Unresectable) or Stage IV Melanoma Progressing Post Prior Systemic Treatment Containing an Anti CTLA-4 Monoclonal Antibody (Checkmate 168: CHECKpoint Pathway for nivoluMAb Clinical Trial Evaluation 168)
Brief Title: Expanded Access Program With Nivolumab to Treat Melanoma
Acronym: Checkmate 168
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-168
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Stage III (Unresectable) or Stage IV Advanced Melanoma
MeSH Terms: interventions — Nivolumab

INTERVENTIONS:
Drug: Nivolumab

SUMMARY:
The purpose of this program is to provide treatment with nivolumab to subjects with Stage III or Stage IV advanced melanoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* ECOG Performance Status of 0-1
* Histologically confirmed malignant melanoma
* Progressed on or after treatment with an anti-CTLA4

Exclusion Criteria:

* Active brain metastases
* Life Expectancy <6 weeks
* Subjects who received prior therapy targeting T-cell costimulation or checkpoint pathways except for Anti CTLA-4 therapy
* Subjects with autoimmune disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2014-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (67):
- United States (23):
  - Local Institution, Mobile, Alabama
  - Southern Cancer Center Pc, Mobile, Alabama
  - Local Institution, Encinitas, California
  - Local Institution, Washington D.C., District of Columbia
  - Lynn Cancer Institute At Boca Raton Regional Hospital, Boca Raton, Florida
  - Cancer Specialists Of North Florida, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Oncology Hematology Associates Of Sw In, Newburgh, Indiana
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Lutherville, Maryland
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - Mid Ohio Oncology/Hematology, Inc,Dba, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - St. Luke'S Hospital, Bethlehem, Pennsylvania
  - The Jones Clinic, Pc, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Argentina (7):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Caba
- Brazil (16):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Brasília, Federal District
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Jd. Petropolis-Londrina, Paraná
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Passo Fundo, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Florianópolis, Santa Catarina
  - Local Institution, Itajaí, Santa Catarina
  - Local Institution, Barretos, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, Ribeirão Preto, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (16):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, North Vancouver, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Moncton, New Brunswick
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Colombia (3):
  - Local Institution, Bogotá
  - Local Institution, Cali
  - Local Institution, Medellín
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Lima

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx